CLINICAL TRIAL: NCT07368881
Title: Fast Food Online Delivery Purchase Behaviour in the Presence and Absence of Price-based Incentives
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Liverpool John Moores University (Other); University of Bristol (Other); Economic and Social Research Council, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pizza promotions study; ES/W007932/1 (Other Grant/Funding Number: Economic and Social Research Council)
Record Dates: First submitted 2026-01-20; First posted 2026-01-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Food Purchases; Eating Behaviour
Keywords: Obesity; Food pricing; Price promotions
MeSH Terms: conditions — Feeding Behavior; Obesity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two conditions
Who Masked: Participant, Investigator
Masking Description: Participants and researchers will not know the group to which individuals have been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control condition (Other): Participants will choose from a food menu with regular pricing, and three price-based incentives present (value pricing, bulk-buy incentives, and price reductions).
  Interventions: Behavioral: Control
- Experimental condition (Experimental): Participants will choose from a menu with no price-based incentives present.
  Interventions: Behavioral: Experimental

INTERVENTIONS:
Behavioral: Experimental — Food menus will provided with all three types of price promotions removed
  Arms: Experimental condition
Behavioral: Control — Participants will be asked to select a meal from a pizza outlet with all price-based incentives present (value pricing, price reductions, bulk-buy incentives).
  Arms: Control condition

SUMMARY:
Consumption of out-of-home (OOH) food is associated with significantly greater energy and less-healthy nutrient (i.e. fats, salt and sugar) intake. The price of food is a key consideration of food choice, particularly for individuals of lower socioeconomic position (SEP). Little research to date has examined the causal effect of removing price-based incentives on purchasing behaviour in OOH food settings. One online randomised controlled trial explored the effect of removing three types of price-based incentives individually and in combination, on food choice through a virtual food delivery platform. This study found that energy selection was 7-8% lower when price incentives were removed. While not statistically significant, Bayes factors indicted that data comparing control vs "all promotions removed" conditions were inconclusive (BF10 = 0.55) and therefore could not provide support for the alternative or null hypotheses. A limitation of this study is that the outcome was hypothetical food choice. As participants would not pay for or receive their selected meals, the prices of foods may have been less salient, thus reducing the potential for impact. In the present study, exploring real-world consumer behaviour (as opposed to hypothetical choice) will better determine the potential impact of removing price-based incentives in the OOH food sector.

DETAILED DESCRIPTION:
See attached study protocol for detailed information

ELIGIBILITY:
Inclusion Criteria:

* Able to order and pay for a takeaway pizza for delivery today or tomorrow
* Currently reside in select postcode areas

  * Manchester (M13 store): M1, M2, M3, M4, M5, M11, M12, M13, M14, M15, M16, M18, M19
  * Liverpool (L3 store): L1, L2, L3, L4, L5, L6, L8, L13, L15
  * Birmingham (B27 store): B9, B10, B11, B12, B13, B25, B26, B27, B28, B33, B90, B91, B92
* Over the age of 18 years
* Report having used food delivery services in the last year

Exclusion Criteria:

* Partaking in a fast or other restrictive eating (e.g. for religious or health reasons) at time of participation
* A previous eating disorder diagnosis
* Currently on appetite-suppressing medication
* Dietary restrictions/intolerances including:

  * Gluten-free
  * Dairy-free
  * Sugar-free

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Energy consumed per household member | The morning after food orders are placed.
  Main participants will select a food order on behalf of their household. The day after receiving their food order, all participants will be asked to estimate the amount of each ordered item that they ate. This information will be used to estimate energy consumed by each household member.

SECONDARY OUTCOMES:
Total monetary spend per household member | Immediately after food choice
  Participants will select their food order. The total monetary value of the food order will be divided by the number of reported household members to get a value of monetary spend per household member.
Energy content per household member | Immediately after food choice
  Participants will select their food order. The total energy content of the food order will be divided by the number of reported household members to get a value of energy content per household member.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liverpool, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Study data (anonymised) will be shared on the Open Science Framework (OSF)
Supporting Information: Study Protocol, SAP
Time Frame: On publication, indefinitely
Access Criteria: Open website
URL: https://osf.io/xeqpc/overview

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2026-01-19): https://cdn.clinicaltrials.gov/large-docs/81/NCT07368881/Prot_SAP_ICF_000.pdf